CLINICAL TRIAL: NCT06820021
Title: The Effects of a Strength-based Tailored-Exercise Program at Home (STEP@Home) on Health Outcomes of Geriatric Patients at Risk of Hospitalization-associated Functional Decline: A Sequential Mixed-method Study
Brief Title: Strength-based Tailored-Exercise Program at Home for Geriatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: STEP@Home full trial
Record Dates: First submitted 2025-01-27; First posted 2025-02-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-06

CONDITIONS: Frailty; Geriatrics
Keywords: Strength-based Tailored-Exercise Program; geriatric care; Hospitalization-associated functional decline; health aging; functional outcome; post-discharge period
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: One research assistant who is blinded to the subjects' group status will measure the outcome variables at the three post-test endpoints (i.e., weeks 12 [T1]. 20 [T2], and 32 [T3]).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The 20-week STEP@Home is a multi-component exercise training program designed to recondition the functional status of older adults in the post-discharge period and to develop long-term exercise engagement. The content is developed based on the recommendations from a scope review and the Vivifrail exercise guideline on home-based exercise for older adults , with expert input from the research team including geriatricians in frailty management, exercise physiologist, nursing academicians in aged care research. Three design characteristics, including an empowerment approach (Funnell & Anderson, 2004), lifestyle-integrated functional exercises (Weber et al., 2018), and an optimized tele-platform, are incorporated into the exercise program to enhance such therapeutic benefit.
  Interventions: Other: Strength-based Tailored-Exercise Program at Home (STEP@Home)
- Control group (Other): The control group will receive a general education delivered by the RA during the first home visit, including general post-discharge knowledge related to frailty, nutrition, mental health, and sleep hygiene, all information are publicly accessible no explicit information related to exercise or physical activity will be included. Five monthly telephone calls will be made to record the information related to the general health of the client at week 4th , 8th, 12th ,16th, and 20th. The RA will make home visit for data collection at 12th, 20th and 32nd week endpoints.
  The RA will also review the post-discharge planning of the client and record information about referral to any social and health care service. The controls will receive a HK$50 supermarket coupon as incentive, and the same will be applied to the intervention group.
  Interventions: Other: Physical activity education

INTERVENTIONS:
Other: Strength-based Tailored-Exercise Program at Home (STEP@Home) — The 20-week STEP@Home is a multi-component exercise training program designed to recondition the functional status of older adults in the post-discharge period and to develop long-term exercise engagement. The content is developed based on the recommendations from a scope review and the Vivifrail exercise guideline on home-based exercise for older adults , with expert input from the research team including geriatricians in frailty management, exercise physiologist, nursing academicians in aged care research. Three design characteristics, including an empowerment approach (Funnell & Anderson, 2004), lifestyle-integrated functional exercises (Weber et al., 2018), and an optimized tele-platform, are incorporated into the exercise program to enhance such therapeutic benefit.
  Arms: Intervention group
Other: Physical activity education — The control group will receive a general education delivered by the RA during the first home visit, including general post-discharge knowledge related to frailty, nutrition, mental health, and sleep hygiene, all information are publicly accessible no explicit information related to exercise or physical activity will be included. Five monthly telephone calls will be made to record the information related to the general health of the client at week 4th , 8th, 12th ,16th, and 20th. The RA will make home visit for data collection at 12th, 20th and 32nd week endpoints.
  The RA will also review the post-discharge planning of the client and record information about referral to any social and health care service. The controls will receive a HK$50 supermarket coupon as incentive, and the same will be applied to the intervention group.
  Arms: Control group

SUMMARY:
This study focuses on the "Strength-based Tailored-Exercise Program at Home (STEP@Home)" aimed at improving health outcomes for geriatric patients at risk of hospitalization-associated functional decline. It is a sequential mixed-method study that combines quantitative and qualitative approaches.

DETAILED DESCRIPTION:
This is a sequential mixed-method study, including a multi-site randomized controlled trial to evaluate the effects of the 20-week STEP@Home program and a subsequent descriptive qualitative study to explore the subjects' experience of program engagement. An overview of the timeline is given in Figure 1. Block randomization with block sizes of 4, 8, and 12, using a restricted shuffled approach with a computer-generated random sequence, will randomly allocate the subjects to receive either STEP@Home or physical activity education at a 1:1 ratio.to develop the STEP@Home intervention, integrating a strength-based, tailored exercise regimen for elderly patients post-hospital discharge. It addresses hospitalization-associated functional decline (HAFD) by engaging patients in sustainable self-practice of physical exercises at home. The study employs empowerment strategies, lifestyle-integrated functional exercises, and optimized tele-platform use to maximize therapeutic benefits. By focusing on empowering patients through sustainable self-practice of physical exercises at home, it aims to enhance physical functions and improve health-related quality of life. The study also has significant real-world implications, potentially offering a scalable, effective solution for the broader geriatric population to manage HAFD, thereby reducing healthcare costs and improving overall well-being. The research intends to assess the program's impact on physical functions and health-related quality of life, utilizing a sequential mixed-method approach for a comprehensive evaluation.

ELIGIBILITY:
Inclusion Criteria:

* i) aged 60 or above
* ii) has an acute hospitalization and the length of hospital stay is of ≥ 2 days2,
* iii) has risk of functional decline in 3 months following hospitalization as measured by the Screening for High-Risk Patients (SHERPA) score of >3.5. SHERPA is a brief measure to identify the high risk by screening for the risk factors, including old age, poor health perception, IADL dysfunction, mild cognitive impairment and fall in the previous year.
* iv) discharged home without any referral for exercise-based rehabilitation
* v) has a Smartphone to access video calls
* vi) consented to participate.

Exclusion Criteria:

* i) admitted with a disabling condition leading to significant functional loss such as stroke,)
* ii) bed-bound or chair bound
* iii) with conditions contradictory to exercise training (e.g., acute muscular-skeletal problem, acute and unstable cardio-respiratory disease, etc),
* iv) engaging in moderate or vigorous exercise (>60min/week) in the past 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
The Short Physical Performance Battery (SPPB) | will be measured at baseline (T0) before randomization and at the 12th (T1), 20th (T2), and 32nd (T3)
  It measures the physical functioning. It combines a balance test, gait velocity, and chair stand to reflect the functional capacity of older adults . Its score ranges from 0-12 in an ascending trend toward increased functional status. The minimal clinically important difference (MCID) is 1.0 for the risk of disability and mortality .The SPPB has good predictive validity against functional decline, rehospitalization and mortality in older adults.

SECONDARY OUTCOMES:
The 11-item Edmonton Frail Scale（EFS） | It will be measured at baseline (T0) before randomization and at the 12th (T1), 20th (T2), and 32nd (T3)
  It measures the level of frailty by positioning an individual on the spectrum of frailty through a multidimensional assessment (Hilmer et al., 2009). It allows a more comprehensive outcome evaluation, especially some of its domains, including cognition, mood, nutritional status, functional independence, and performance, which were responsive to post-discharge exercise training among older adults.18 Its brevity only requires 5-10 minutes for completion, and the EFS has good reliability, stability, and criterion validity in older Chinese adults
The Life Space Assessment (LSA-C) | It will be measured at baseline (T0) before randomization and at the 12th (T1), 20th (T2), and 32nd (T3)
  It measures physical function in terms of mobility level in everyday activities. It assesses mobility level at five life-space levels in the past 4 weeks: i) living room other than the bedroom, ii) outside the house, iii) the neighborhood (within 800m of home), iv) outside the neighborhood (within 8km) and v) outside the town (beyond 16km). Example locations representing various distances from subjects' homes will be provided to facilitate the responses. The reliability of LSA-C is 0.88, with good criterion and construct validity
EuroQoL-5D-5L will assess HRQoL | It will be measured at baseline (T0) before randomization and at the 12th (T1), 20th (T2), and 32nd (T3)
  It comprises a 5-level response set (5-L), including mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a 0-100 visual analogue scale to measure perceived health. The EuroQoL-5D-5L is more discriminative than the conventional 3L version for, with a Cronbach's alpha of 0.86
qualitative data collection | It will be conducted at T2
  As for the qualitative data collection, the interviews will be conducted for the 30 subjects recruited through purposive sampling. Broad, open-ended questions will guide the semi-structured interview, which focuses on the perceived effects of STEP@Home on functional and health status, how it works (if any) or not works, challenges of implementation, and concerns of longer-term exercise engagement. The findings will enhance the interpretation of the quantitative outcome-based evaluation.
Hospital Admission and Emergency Department Attendance | It will be collected at baseline (T0), and 1 year
  Hospital admission and Emergency Department Attendance data including number of attendance, length of stay, and major diagnosis will be collected as health-related outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- the University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tseng YC, Gau BS, Lou MF. Validation of the Chinese version of the Life-Space Assessment in community-dwelling older adults. Geriatr Nurs. 2020 Jul-Aug;41(4):381-386. doi: 10.1016/j.gerinurse.2019.11.014. Epub 2019 Dec 7. PMID 31818502
- [Result] Sunde S, Hesseberg K, Skelton DA, Ranhoff AH, Pripp AH, Aaronaes M, Brovold T. Effects of a multicomponent high intensity exercise program on physical function and health-related quality of life in older adults with or at risk of mobility disability after discharge from hospital: a randomised controlled trial. BMC Geriatr. 2020 Nov 11;20(1):464. doi: 10.1186/s12877-020-01829-9. PMID 33176703
- [Result] Lee JS, Auyeung TW, Leung J, Kwok T, Woo J. Transitions in frailty states among community-living older adults and their associated factors. J Am Med Dir Assoc. 2014 Apr;15(4):281-6. doi: 10.1016/j.jamda.2013.12.002. Epub 2014 Feb 16. PMID 24534517
- [Result] Izquierdo M. [Multicomponent physical exercise program: Vivifrail]. Nutr Hosp. 2019 Jul 1;36(Spec No2):50-56. doi: 10.20960/nh.02680. Spanish. PMID 31189323
- [Result] Guralnik JM, Winograd CH. Physical performance measures in the assessment of older persons. Aging (Milano). 1994 Oct;6(5):303-5. doi: 10.1007/BF03324256. No abstract available. PMID 7893776
- [Result] Ashworth NL, Chad KE, Harrison EL, Reeder BA, Marshall SC. Home versus center based physical activity programs in older adults. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD004017. doi: 10.1002/14651858.CD004017.pub2. PMID 15674925
- [Result] Zisberg A, Shadmi E, Sinoff G, Gur-Yaish N, Srulovici E, Admi H. Low mobility during hospitalization and functional decline in older adults. J Am Geriatr Soc. 2011 Feb;59(2):266-73. doi: 10.1111/j.1532-5415.2010.03276.x. PMID 21314647
- [Result] Weber M, Belala N, Clemson L, Boulton E, Hawley-Hague H, Becker C, Schwenk M. Feasibility and Effectiveness of Intervention Programmes Integrating Functional Exercise into Daily Life of Older Adults: A Systematic Review. Gerontology. 2018;64(2):172-187. doi: 10.1159/000479965. Epub 2017 Sep 15. PMID 28910814
- [Result] Tavares JPA, Nunes LANV, Gracio JCG. Hospitalized older adult: predictors of functional decline. Rev Lat Am Enfermagem. 2021 Jan 8;29:e3399. doi: 10.1590/1518-8345.3612.3399. eCollection 2021. PMID 33439951
- [Result] McCullagh R, O'Connell E, O'Meara S, Dahly D, O'Reilly E, O'Connor K, Horgan NF, Timmons S. Augmented exercise in hospital improves physical performance and reduces negative post hospitalization events: a randomized controlled trial. BMC Geriatr. 2020 Feb 7;20(1):46. doi: 10.1186/s12877-020-1436-0. PMID 32033532
- [Result] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Saez de Asteasu ML, Lucia A, Galbete A, Garcia-Baztan A, Alonso-Renedo J, Gonzalez-Glaria B, Gonzalo-Lazaro M, Apezteguia Iraizoz I, Gutierrez-Valencia M, Rodriguez-Manas L, Izquierdo M. Effect of Exercise Intervention on Functional Decline in Very Elderly Patients During Acute Hospitalization: A Randomized Clinical Trial. JAMA Intern Med. 2019 Jan 1;179(1):28-36. doi: 10.1001/jamainternmed.2018.4869. PMID 30419096
- [Result] Loyd C, Markland AD, Zhang Y, Fowler M, Harper S, Wright NC, Carter CS, Buford TW, Smith CH, Kennedy R, Brown CJ. Prevalence of Hospital-Associated Disability in Older Adults: A Meta-analysis. J Am Med Dir Assoc. 2020 Apr;21(4):455-461.e5. doi: 10.1016/j.jamda.2019.09.015. Epub 2019 Nov 14. PMID 31734122
- [Result] Hilmer SN, Perera V, Mitchell S, Murnion BP, Dent J, Bajorek B, Matthews S, Rolfson DB. The assessment of frailty in older people in acute care. Australas J Ageing. 2009 Dec;28(4):182-8. doi: 10.1111/j.1741-6612.2009.00367.x. PMID 19951339
- [Result] Greysen SR, Stijacic Cenzer I, Auerbach AD, Covinsky KE. Functional impairment and hospital readmission in Medicare seniors. JAMA Intern Med. 2015 Apr;175(4):559-65. doi: 10.1001/jamainternmed.2014.7756. PMID 25642907
- [Result] Geyskens L, Jeuris A, Deschodt M, Van Grootven B, Gielen E, Flamaing J. Patient-related risk factors for in-hospital functional decline in older adults: A systematic review and meta-analysis. Age Ageing. 2022 Feb 2;51(2):afac007. doi: 10.1093/ageing/afac007. PMID 35165688
- [Result] de Foubert M, Cummins H, McCullagh R, Brueton V, Naughton C. Systematic review of interventions targeting fundamental care to reduce hospital-associated decline in older patients. J Adv Nurs. 2021 Dec;77(12):4661-4678. doi: 10.1111/jan.14954. Epub 2021 Jul 9. PMID 34240755
- [Result] Cornette P, Swine C, Malhomme B, Gillet JB, Meert P, D'Hoore W. Early evaluation of the risk of functional decline following hospitalization of older patients: development of a predictive tool. Eur J Public Health. 2006 Apr;16(2):203-8. doi: 10.1093/eurpub/cki054. Epub 2005 Aug 2. PMID 16076854
- [Result] Clegg AP, Barber SE, Young JB, Forster A, Iliffe SJ. Do home-based exercise interventions improve outcomes for frail older people? Findings from a systematic review. Rev Clin Gerontol. 2012 Feb;22(1):68-78. doi: 10.1017/S0959259811000165. Epub 2012 Aug 24. PMID 27226701
- [Result] Boyd CM, Landefeld CS, Counsell SR, Palmer RM, Fortinsky RH, Kresevic D, Burant C, Covinsky KE. Recovery of activities of daily living in older adults after hospitalization for acute medical illness. J Am Geriatr Soc. 2008 Dec;56(12):2171-9. doi: 10.1111/j.1532-5415.2008.02023.x. PMID 19093915
- [Result] Bilbao A, Garcia-Perez L, Arenaza JC, Garcia I, Ariza-Cardiel G, Trujillo-Martin E, Forjaz MJ, Martin-Fernandez J. Psychometric properties of the EQ-5D-5L in patients with hip or knee osteoarthritis: reliability, validity and responsiveness. Qual Life Res. 2018 Nov;27(11):2897-2908. doi: 10.1007/s11136-018-1929-x. Epub 2018 Jul 5. PMID 29978346
- [Result] Admi H, Shadmi E, Baruch H, Zisberg A. From research to reality: minimizing the effects of hospitalization on older adults. Rambam Maimonides Med J. 2015 Apr 29;6(2):e0017. doi: 10.5041/RMMJ.10201. eCollection 2015 Apr. PMID 25973269

DOCUMENTS (1):
  • Informed Consent Form (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT06820021/ICF_000.pdf